CLINICAL TRIAL: NCT03543085
Title: A Single-arm, Open Label, Single Center, Prospective Study of Ultra-high Frequency (500 KHz) Spinal Cord Stimulation for Treatment of Chronic Back Pain or Lower Limb Pain
Brief Title: Ultra-high Frequency (500 KHz) Spinal Cord Stimulation for Treatment of Chronic Back Pain or Lower Limb Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GiMer Medical (Industry)
Collaborators: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PT1710001
Record Dates: First submitted 2018-05-18; First posted 2018-06-01 (Actual); Results first posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Pain, Chronic; Pain, Back; Pain, Radiating
MeSH Terms: conditions — Chronic Pain; Back Pain; Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrahigh Frequency (500 KHz) Stimulation (Experimental): This study is a prospective, single-arm, open label, single center to confirm the effectiveness and safety of an ultrahigh frequency spinal cord stimulation in patients with chronic back pain or lower limb pain.
  Interventions: Device: GiMer Medical MN 1000 External Stimulator

INTERVENTIONS:
Device: GiMer Medical MN 1000 External Stimulator — Trial stimulator (GiMer Medical Model 1000 External Stimulator) to generate pulsed ultrahigh frequency (>200KHz) electrical stimulation, delivered via lead in epidural space, in treating pain. Similar with current market available Spinal Cord Stimulators but with a higher stimulation frequency (hundred KHz) range.

SUMMARY:
This study is a prospective, single-arm, open label, single center to confirm the effectiveness and safety of an ultra-high frequency (500 KHz) spinal cord stimulation in patients with chronic back pain or lower limb pain.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, open label, single center to confirm the effectiveness and safety of an ultra-high frequency (500 KHz) spinal cord stimulation in patients with chronic back pain or lower limb pain. The trial length is 14 days. Patients will be given ultrahigh frequency pulse stimulation, up to 3 times in every 24 hours, and VAS will be obtained at least once a day. Compared to previous study conducted last year, patient can now have two lead implant sites for different pain locations. The electrode implantation site will be epidural space instead of Dorsal Root Ganglion (DRG).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≧20 and ≦75
2. Have a symptom of back or lower limb pain with a diagnosis related to spinal lesion, herniated disc, nerve injury, stenosis, failed back surgery syndrome (FBSS), complex regional pain syndrome (CRPS) or ischemic lower limb pain and have pain history of >6 months.
3. Have an average pain score >5 by Visual Analogue Scale (VAS) on inclusion.
4. Has failed to achieve adequate pain relief from prior pharmacologic treatments.
5. In the judgement of the investigator, the subject is an appropriate candidate for the trial procedure.
6. The subject is willing and able to comply with the procedure and requirements of this trial.
7. The participant is able to understand and provide informed consent, and has signed their written informed consent in accordance with Institutional Review Board (IRB) requirements.

Exclusion Criteria:

1. Have evidence of a mental or psychological condition that affects pain perception and has difficulty/disability performing objective pain assessment, or have previously failed mental or psychological assessments administered by a psychiatrist that may be deemed to indicate the subject's lack of suitability for participation in this study.
2. Subject has exhibited unstable pain condition within the past 30 days as interviewed by Investigator.
3. Be on anticoagulant medication with International Normalized Ratio (INR) >1.5 or platelet count less than 100,000/μL, peripheral vascular diseases (PVDs), visceral pain or uncontrolled Diabetes mellitus (DM).
4. Has had corticosteroid therapy at an intended site of stimulation within the past 30 days.
5. Pain medication(s) dosages(s) are not stable for at least 30 days at investigator's discretion.
6. Currently has an active implantable device including International Classification of Diseases (ICD), pacemaker, spinal cord stimulator or intrathecal drug pump or subject requires magnetic resonance imaging (MRIs) or diathermy.
7. Have a current diagnosis of cancer with active symptoms.
8. Have a known terminal illness with life expectancy less than one year.
9. Have a systematic or local infection, which may increase study risk.
10. Currently has an indwelling device that may pose an increased risk of infection.
11. Be pregnant or breast feeding.
12. Have a medical history of drug or alcohol addiction within the past 2 years.
13. Participation in any investigational study in the last 30 days or current enrollment in any trial.
14. Be currently involved in an injury claim law suit or medically related litigation, including workers compensation.
15. Be a prisoner.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-10-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultrahigh Frequency (500 KHz) Stimulation
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ultrahigh Frequency (500 KHz) Stimulation
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 43.5 [24.9 to 65.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Analog Score From Baseline to Day 14
Description: To assess the analgesic effectiveness of ultra-high frequency spinal cord stimulation, as measured by Visual Analogue Scale (VAS, score min 0 no pain to max 10 worst pain) compared to baseline.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ultrahigh Frequency (500 KHz) Stimulation
Number analyzed (Participants) | 10
score on a scale | -5.1 (2.3)

2. Primary Outcome: Record Incidence of Adverse Events
Description: To evaluate safety of ultra-high frequency spinal cord stimulation by identifying the incidence rate of adverse events (AEs) and serious adverse events (SAEs) during the trial
Time Frame: 14 days
Measure: Number; unit: events
Arm/Group | Ultrahigh Frequency (500 KHz) Stimulation
Number analyzed (Participants) | 10
events | 16

3. Secondary Outcome: The Brief Pain Inventory (BPI)
Description: The change from baseline in functionality using the BPI evaluations
Time Frame: 14 days
Reporting Status: Not Posted

4. Secondary Outcome: Incidence of Stimulation-induced Paresthesia
Description: To determine the presence or absence of stimulation-induced paresthesia.
Time Frame: 14 days
Reporting Status: Not Posted

5. Secondary Outcome: Pain Relief Medication Consumption
Description: Amount of pain medication consumption, including Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) and weak opioids, compared to baseline
Time Frame: 14 days
Reporting Status: Not Posted

6. Secondary Outcome: Oswestry Low Back Pain Disability Questionnaire (ODI)
Description: The change from baseline in functionality using the ODI evaluations
Time Frame: 14 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 14 days from baseline
Arm/Group | Ultrahigh Frequency (500 KHz) Stimulation
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ultrahigh Frequency (500 KHz) Stimulation (N=10)
Incision site pain (Injury, poisoning and procedural complications) | 7 (7)
headache (Nervous system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/85/NCT03543085/Prot_SAP_000.pdf